CLINICAL TRIAL: NCT01269671
Title: Efficacy of Combination Therapy vs Placebo for Pediatric Functional Abdominal Pain
Acronym: FAP
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI has left institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Adrian Miranda, MD (Associate Professor), Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHW 10/102
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Functional Abdominal Pain; Irritable Bowel Syndrome; Functional Dyspepsia
Keywords: Functional Abdominal Pain; Irritable Bowel Syndrome; IBS; Functional Dyspepsia; Melatonin; Simethicone; Peppermint Oil; mentharil; functional bowel disorders; quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Melatonin; peppermint oil; Simethicone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin, Peppermint Oil, Simethicone (Experimental)
  Interventions: Drug: Melatonin, Peppermint Oil (mentharil), and Simethicone
- Sugar pill (Placebo Comparator)
  Interventions: Other: Sugar pill

INTERVENTIONS:
Drug: Melatonin, Peppermint Oil (mentharil), and Simethicone — Dosing will be dependent on patient's age during time of enrollment. Patients 8-12 years of age will receive Melatonin 3mg tab at night, Peppermint oil 1 capsule (0.2ml) 30-60 minutes prior to meal twice daily, and Simethicone 80mg tab 30-60 minutes prior to meal twice daily. Patients 13-18 years of age will receive Melatonin 3mg tab at night, Peppermint oil 2 capsules (0.4ml) 30-60 minutes prior to meal twice daily, and Simethicone tab 125mg 30-60 minutes prior to meal twice daily
  Arms: Melatonin, Peppermint Oil, Simethicone
Other: Sugar pill — Patients in the placebo group will receive one placebo tab to be taken at night, one placebo capsule to be taken 30-60 minutes prior to meal twice daily, and one placebo tab to be taken 30-60 minutes prior to meal twice daily.
  Arms: Sugar pill

SUMMARY:
IND application was submitted to FDA on November 17th.

ELIGIBILITY:
Inclusion Criteria: To participate in this study, the child/teen must be a patient of the FAP Clinic/GI Clinic in the Division of Gastroenterology at the Children's Hospital of Wisconsin, and have a parent or legal guardian who is willing to participate. Children aged 8-18 years will be eligible for inclusion in the study.

Exclusion Criteria: Children or parents who are non-English speaking, or parents and/or children with cognitive delay that precludes comprehension and completion of questionnaires will be excluded from participating in this registry.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | 8 weeks
  To evaluate the efficacy of the treatment combination of Melatonin, Peppermint Oil, and Simethicone in releiving the symptoms of pain in Irritable Bowel Syndrome, Functional Abdominal Pain, and Functional Dyspepsia compared to treatment outcomes to placebo.
Quality of Life | 8 weeks
  To evaluate improvement in quality of life in children treated with combination therapy versus placebo.
Anxiety Affects | 8 weeks
  To determine if patient anxiety affects treatment outcomes in patients with functional bowel disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Miranda, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Saps M, Seshadri R, Sztainberg M, Schaffer G, Marshall BM, Di Lorenzo C. A prospective school-based study of abdominal pain and other common somatic complaints in children. J Pediatr. 2009 Mar;154(3):322-6. doi: 10.1016/j.jpeds.2008.09.047. Epub 2008 Nov 28. PMID 19038403
- [Background] Youssef NN, Murphy TG, Langseder AL, Rosh JR. Quality of life for children with functional abdominal pain: a comparison study of patients' and parents' perceptions. Pediatrics. 2006 Jan;117(1):54-9. doi: 10.1542/peds.2005-0114. PMID 16396860
- [Background] Schurman JV, Danda CE, Friesen CA, Hyman PE, Simon SD, Cocjin JT. Variations in psychological profile among children with recurrent abdominal pain. J Clin Psychol Med Settings. 2008 Sep;15(3):241-51. doi: 10.1007/s10880-008-9120-0. Epub 2008 Jul 25. PMID 19104969
- [Background] White KS, Farrell AD. Anxiety and psychosocial stress as predictors of headache and abdominal pain in urban early adolescents. J Pediatr Psychol. 2006 Jul;31(6):582-96. doi: 10.1093/jpepsy/jsj050. Epub 2005 Jul 27. PMID 16049263
- [Background] Saps M, Youssef N, Miranda A, Nurko S, Hyman P, Cocjin J, Di Lorenzo C. Multicenter, randomized, placebo-controlled trial of amitriptyline in children with functional gastrointestinal disorders. Gastroenterology. 2009 Oct;137(4):1261-9. doi: 10.1053/j.gastro.2009.06.060. Epub 2009 Jul 31. PMID 19596010
- [Background] Klupinska G, Poplawski T, Drzewoski J, Harasiuk A, Reiter RJ, Blasiak J, Chojnacki J. Therapeutic effect of melatonin in patients with functional dyspepsia. J Clin Gastroenterol. 2007 Mar;41(3):270-4. doi: 10.1097/MCG.0b013e318031457a. PMID 17426465
- [Background] Song GH, Leng PH, Gwee KA, Moochhala SM, Ho KY. Melatonin improves abdominal pain in irritable bowel syndrome patients who have sleep disturbances: a randomised, double blind, placebo controlled study. Gut. 2005 Oct;54(10):1402-7. doi: 10.1136/gut.2004.062034. Epub 2005 May 24. PMID 15914575
- [Background] Mickle A, Sood M, Zhang Z, Shahmohammadi G, Sengupta JN, Miranda A. Antinociceptive effects of melatonin in a rat model of post-inflammatory visceral hyperalgesia: a centrally mediated process. Pain. 2010 Jun;149(3):555-564. doi: 10.1016/j.pain.2010.03.030. Epub 2010 Apr 21. PMID 20413219
- [Background] Kline RM, Kline JJ, Di Palma J, Barbero GJ. Enteric-coated, pH-dependent peppermint oil capsules for the treatment of irritable bowel syndrome in children. J Pediatr. 2001 Jan;138(1):125-8. doi: 10.1067/mpd.2001.109606. PMID 11148527
- [Background] Voepel-Lewis TD, Malviya S, Burke C, D'Agostino R, Hadden SM, Siewert M, Tait AR. Evaluation of simethicone for the treatment of postoperative abdominal discomfort in infants. J Clin Anesth. 1998 Mar;10(2):91-4. doi: 10.1016/s0952-8180(97)00249-3. PMID 9524891
- [Background] Kaplan MA, Prior MJ, Ash RR, McKonly KI, Helzner EC, Nelson EB. Loperamide-simethicone vs loperamide alone, simethicone alone, and placebo in the treatment of acute diarrhea with gas-related abdominal discomfort. A randomized controlled trial. Arch Fam Med. 1999 May-Jun;8(3):243-8. doi: 10.1001/archfami.8.3.243. PMID 10333820